CLINICAL TRIAL: NCT04650438
Title: Sleep and Creativity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not start due to COVID-19 pandemic.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018-01578
Record Dates: First submitted 2020-11-19; First posted 2020-12-02 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Creativity Performance in Healthy Subjects
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, cross-over trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-creativity (Experimental): Here participants are allocated to the high-creativity group. Resting state EEG will be measured pre- and post-TMS and participants' creative performance will be measured by means of a creativity test battery.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) over the left inferior frontal gyrus (IFG); Device: Transcranial Magnetic Stimulation (TMS) over the left inferior parietal lobule (IPL)
- Low-creativity (Experimental): Here participants are allocated to the low-creativity group. Resting state EEG will be measured pre- and post-TMS and participants' creative performance will be measured by means of a creativity test battery.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) over the left inferior frontal gyrus (IFG); Device: Transcranial Magnetic Stimulation (TMS) over the left inferior parietal lobule (IPL)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) over the left inferior frontal gyrus (IFG) — MagPro X100, with MagPro software version 7.1; connected to a figure-of-eight coil (MC-B70) or a circular coil (MC-125). The device is CE marked and bears an ISO 13485 certificate complying with good manufacturing practice. Continuous theta burst stimulation protocol will be applied.
Device: Transcranial Magnetic Stimulation (TMS) over the left inferior parietal lobule (IPL) — MagPro X100, with MagPro software version 7.1; connected to a figure-of-eight coil (MC-B70) or a circular coil (MC-125). The device is CE marked and bears an ISO 13485 certificate complying with good manufacturing practice. Continuous theta burst stimulation protocol will be applied.

SUMMARY:
Creativity is a complex neuro-psycho-philosophical phenomenon that is difficult to define. Neurocognitive models of creativity suggest that creativity is associated with the activity of a distributed, bilateral fronto-temporal and parietal network. Therefore, a modulation of frontal activity is necessary to allow a certain degree of "controlled disinhibition", which seems to be necessary for creative thinking. In addition, a modulation of the lower parietal lobe (IPL) might allow targeting the brain regions responsible for idea generation.

This project will investigate the application of transcranial magnetic stimulation (TMS) with the intent of modulating creativity performance of healthy subjects. Resting state electroencephalography (EEG) that will be acquired pre- and post-TMS and participants' creative performance will be measured.

Perspectives include a better understanding of the differences between high- and low-creativity groups, as measured by a creativity test battery, in their response to TMS. Additional perspectives are whether there are differences in creativity performance depending on the stimulation location.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age between 18 and 70 years
* Neurologically healthy, i.e., with no documented or present neurological disease or brain injury
* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* Any instable medical condition, in particular epilepsy (past or pre-sent, including seizures or febrile convulsions)
* Any surgical intervention to the brain
* Implanted medical devices (e.g., cochlear implants, infusion pumps, neurostimulators, pacemakers)
* Presence of metal in the region of the head (excluding fixed dental implants such as tooth fillings or fixed dental braces)
* Drug or alcohol abuse
* Intake of any medication that is likely to lower seizure threshold
* For female participants: in order to participate in the study, female patients in reproductive age need to take a pregnancy test (a stand-ard urine pregnancy test will be provided).
* Previous enrolment in a creativity study of the same PI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in creativity performance prior- and post-TMS | 2.5 hours
  Change in creativity performance (as expressed by a summary score of single tests from a creativity test battery) prior- and post-TMS in low- and high-creativity groups

SECONDARY OUTCOMES:
Change in creativity performance prior- and post-TMS depending on stimulation location | 2.5 hours
  Change in creativity performance (as expressed by a summary score of single tests from a creativity test battery) prior- and post-TMS depending on the stimulation location (left IFG versus left IPL)

CONTACTS AND LOCATIONS:
Overall Officials: René M. Müri, Prof. Dr., Principal Investigator — Department of Neurology Inselspital, Bern University Hospital; Claudio Bassetti, Prof. Dr., Study Chair — Department of Neurology Inselspital, Bern University Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Beaty RE, Benedek M, Wilkins RW, Jauk E, Fink A, Silvia PJ, Hodges DA, Koschutnig K, Neubauer AC. Creativity and the default network: A functional connectivity analysis of the creative brain at rest. Neuropsychologia. 2014 Nov;64:92-8. doi: 10.1016/j.neuropsychologia.2014.09.019. Epub 2014 Sep 20. PMID 25245940
- [Background] Jung J, Bungert A, Bowtell R, Jackson SR. Vertex Stimulation as a Control Site for Transcranial Magnetic Stimulation: A Concurrent TMS/fMRI Study. Brain Stimul. 2016 Jan-Feb;9(1):58-64. doi: 10.1016/j.brs.2015.09.008. Epub 2015 Sep 25. PMID 26508284
- [Background] Lustenberger C, Boyle MR, Foulser AA, Mellin JM, Frohlich F. Functional role of frontal alpha oscillations in creativity. Cortex. 2015 Jun;67:74-82. doi: 10.1016/j.cortex.2015.03.012. Epub 2015 Apr 1. PMID 25913062
- [Background] Nyffeler T, Wurtz P, Pflugshaupt T, von Wartburg R, Luthi M, Hess CW, Muri RM. One-Hertz transcranial magnetic stimulation over the frontal eye field induces lasting inhibition of saccade triggering. Neuroreport. 2006 Feb 27;17(3):273-5. doi: 10.1097/01.wnr.0000199468.39659.bf. PMID 16462596
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Park HR, Kirk IJ, Waldie KE. Neural correlates of creative thinking and schizotypy. Neuropsychologia. 2015 Jul;73:94-107. doi: 10.1016/j.neuropsychologia.2015.05.007. Epub 2015 May 12. PMID 25979607
- [Background] Vartanian O, Beatty EL, Smith I, Blackler K, Lam Q, Forbes S. One-way traffic: The inferior frontal gyrus controls brain activation in the middle temporal gyrus and inferior parietal lobule during divergent thinking. Neuropsychologia. 2018 Sep;118(Pt A):68-78. doi: 10.1016/j.neuropsychologia.2018.02.024. Epub 2018 Feb 23. PMID 29477840